CLINICAL TRIAL: NCT06802640
Title: Transcutaneous Spinal Cord Electrical Stimulation Combined With Kunming Locomotor Training for the Treatment of Spinal Cord Injury
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kunming Tongren Hospital (Industry)
Responsible Party: Principal Investigator, Hui Zhu, Director, Kunming Tongren Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KunmingTH_HZ_004
Record Dates: First submitted 2025-01-26; First posted 2025-01-31 (Actual); Last update posted 2025-01-31 (Actual); Status verified 2025-01

CONDITIONS: Spinal Cord Injuries
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental)
  Interventions: Combination Product: Transcutaneous spinal cord electrical stimulation and Kunming Locomotor Training
- Group B (Sham Comparator)
  Interventions: Combination Product: Transcutaneous spinal cord electrical stimulation and Kunming Locomotor Training

INTERVENTIONS:
Combination Product: Transcutaneous spinal cord electrical stimulation and Kunming Locomotor Training — Patients will undergo Kunming Locomotor Training along with transcutaneous spinal cord stimulation. . The training is at least 1 hour per day, 5 hours per week, for 6 consecutive months.

SUMMARY:
Spinal cord injury (SCI) is a common and severe traumatic central nervous system injury in clinical practice. Currently, the treatment of SCI remains a worldwide challenge.International studies have confirmed that TSCS is an effective non-invasive technique to activate the body's movement-related circuits. This method utilizes a unique stimulation waveform that is transmitted through electrodes placed on the skin of the spine and spreads through the dorsal roots (DRs) to activate the spinal cord neural circuits.The main objective of this study is to have patients with chronic incomplete (AIS B/C/D) spinal cord injuries wear "transcutaneous spinal cord electrical stimulator " and undergo "Kunming locomotor training" for 6 months, observe the synergistic effects of the two, and evaluate whether this treatment method can improve patients' motor functions.

ELIGIBILITY:
Inclusion Criteria:

* 1. Chronic (≧6 months) paraplegics (T1-T10) with incomplete(AIS B/C/D) spinal cord injury Incomplete aged 16-50 years;
* 2.Subjects must be able to read, understand, and complete the Visual Analogue Scale;
* 3.Subjects voluntarily sign the informed consent form approved by the ethics committee.

Exclusion Criteria:

* 1. Obvious renal, cardiovascular, hepatic, and mental diseases;
* 2.Pregnant or lactating women and women of childbearing age who are unwilling to use contraception;
* 3. Limb contracture deformity;
* 4. Modified Ashworth > Grade 2;
* 5. Unhealed fractures;
* 6. The subject is currently participating in other studies;
* 7. The researcher's opinion is that the subject does not comply with the research protocol and/or is not suitable to participate in this study.

Ages: 16 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 18 (Estimated)
Dates: Start 2025-02-01 (Estimated); Primary Completion 2027-10-31 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline Kunming Locomotor Scale (KLS) at 6 months | Day 0, Month 6
  Scale from minimum (1) to maximum (10), higher scales mean a better outcome.
Change from Baseline 10 Meter Walk Test (10mWT) at 6 months | Day 0, Month 6
  The primary measure obtained from the test is the walking speed, which is calculated by dividing the distance by the time taken to complete the walk.

SECONDARY OUTCOMES:
Change from Baseline Spinal cord injury functional ambulation profile (SCI-FAP) at 6 months | Day 0, Month 6
  Higher scores generally indicate greater independence and better walking ability.
Change from Lower extremity motor score(LEMS) at 6 months | Day 0, Month 6
  a lower score indicates greater motor impairment in the lower extremities

OTHER OUTCOMES:
Change from Walking Index for Spinal Cord Injury (WISCI) at 6 months | Day 0, Month 6
  Higher scores generally indicate greater independence.

IPD SHARING:
Plan to Share IPD: No